CLINICAL TRIAL: NCT02360618
Title: A Window of Opportunity Study to Evaluate the Role of the Combination of Metformin and Simvastatin as a Neoadjuvant Therapy in Invasive Bladder Cancer
Brief Title: Metformin and Simvastatin Use in Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Jonathan Izawa, Urologic Surgeon, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS_1
Record Dates: First submitted 2015-01-13; First posted 2015-02-10 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Metformin; Simvastatin; Combination Therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Metformin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin and Simvastatin Treatment (Experimental): Patients in this group will receive 850 mg of Metformin and 20 mg of Simvastatin daily from the time they are enrolled in the study until the day before their surgery (approximately 12 weeks), in the absence of any safety or tolerability concerns.
  Interventions: Drug: Metformin; Drug: Simvastatin

INTERVENTIONS:
Drug: Metformin — See Group Description
  Other Names: No other names
Drug: Simvastatin — See Group Description
  Other Names: No other names

SUMMARY:
A single arm, single center window of opportunity trial of using a combination of metformin and simvastatin as a neoadjuvant treatment for patients with invasive bladder cancer who are to undergo cystectomy. The study will assess the feasibility of conducting window of opportunity trials in invasive bladder cancer the drug combination's affects on a variety of important clinicopathologic variables.

The goal is to enroll 44 patients within 18 months. An interim analysis will be conducted at 12 months, and the study will be prematurely closed if fewer than 10 patients have been enrolled at that time. Patients will be administered 850mg of metformin twice daily along with 20mg of Simvastatin. Patients will be enrolled following the formal diagnosis of invasive bladder cancer or at first visit following referral to the London Health Sciences Center (LHSC). Patient's will receive metformin and simvastatin from the time of enrollment until the night prior to their operation in the absence of safety or tolerability concerns.

DETAILED DESCRIPTION:
This is a single centre window of opportunity trial. A total of 44 patients with a diagnosis of invasive bladder cancer diagnosed by pathologic evaluation of transurethral resection of bladder tumor (TURBT) specimens and meeting all eligibility criteria will be enrolled in the study. Study participants will receive Metformin 850mg twice daily and simvastatin 20mg once daily until the night before of their scheduled cystectomy, which is a time period which will last approximately 12 weeks or less. Pre-treatment TURBT tissue samples and the Cystectomy post-therapy tissue samples will be analyzed and compared. Samples will be analyzed for cell proliferation markers and to determine whether or not the combination of metformin and simvastatin is able to produce a synergistic effect that will result in the decrease of the growth of these aggressive cancer cells. The anticipated recruitment period will be approximately 18 months. Participants in this study will be asked to attend the following clinic visits for this study:

Baseline Visit:

During this visit, the study doctor will conduct a physical exam and take vital signs as well as height and weight measurements. Blood will also be drawn for analysis and research purposes. Females that are of child bearing potential will have a pregnancy test to confirm that they are not pregnant. Pregnant women will be removed from the study. We will also be collecting blood samples.

Clinic Visits Participants will have follow-up clinic visits or phone interviews scheduled every 4 weeks until the time of their surgery. At least 1 visit will be in person before surgery. At these times they will have blood drawn for analysis, have their medication reviewed, and confirm that they are taking the medication in adherence with the study protocol.

Day of Surgery On the day of surgery, the participants will have their height and weight measured, have blood drawn for analysis and research purposes, and drug compliance will be assessed.

This is a feasibility study, and an interim analysis of enrollment is planned at 12 months after the first patient is enrolled. The trial will be prematurely closed if it fails to enroll 10 patients by the 12 month time point. A preliminary pathological analysis will be performed following the completion of 12 months from the time of study initiation.

In the event that the enrolled patient underwent a TURBT for diagnosis prior to referral, either tissue will be obtained from the peripheral center where the TURBT was performed or they will be consented for repeat TURBT, or withdrawn from the study.

Based upon the documentation at the time of TURBT, an attempt will be made, where possible, to obtain tissue sections from the same tumor contained in the cystectomy sections. Where this is not possible, representative slides will be obtained from another tumor, if available.

Study Objectives The aim of this study is to evaluate feasibility of window of opportunity neoadjuvant trials for invasive bladder cancer in our center, and to determine the effect of the combination of metformin and simvastatin on clinicopathologic markers of drug activity in our patient cohort.

Primary Objectives - Feasibility and Tumor Proliferation Rate The primary endpoint of this trial will be the assessment of the tumor proliferation rate. This will be investigated through the analysis of the change in Ki67 tissue staining between the TURBT tissue samples and the cystectomy tissue.

Marker of cell proliferation;

1. Ki67 staining

   This trial is also designed to establish the framework and evaluate the feasibility of performing neoadjuvant window of opportunity trials using drugs with potential bioactivity against invasive bladder cancer at the London Health Sciences Center. The goal is to accrue 44 patients within 18 months to the trial. A midterm analysis at 12 months will be performed, at which time the trial will be prematurely closed if there have been fewer than 10 patients enrolled.
2. Feasibility - goal to accrue 44 patients in 18 months.

Secondary Objectives This study will assess the rate of grade 3 or higher toxicity as defined by the CTCAE 4.03 (Common Terminology Criteria for Adverse Events). If 41 patients are enrolled and complete the study, the study will have an 85% power at an of 0.05 to detect if the toxicity rate is >20% with an assumed baseline of ≤5%.

1. Toxicity

   The following parameters will be investigated through the analysis of any differences in their tissue staining between the TURBT tissue samples and the cystectomy tissue. This should aid in the delineation of any therapeutic effects of the combination of metformin and simvastatin therapy on urothelial carcinoma (UC).

   Marker of Apoptosis;
2. Terminal deoxynucleotidyl Transferase-mediated deoxy uridine triphosphate (dUTP) nick end labeling (TUNEL) staining

   Phosphoinositide-3 kinase/protein kinase B/mammalian target of rapamycin (PI3K/Akt/mTOR) pathway readouts;
3. p-mTOR staining
4. p-Akt staining
5. survivin

   Metformin stimulates activation;
6. phosphorylated adenosine monophosphate-activated protein kinase (p-AMPK)

   The following parameters will be investigated through the analysis of their tissue staining in the cystectomy sample, as they are assumed to be dependent on the underlying tumor biology and will not be affected by metformin therapy:

   PI3K/Akt/mTOR pathway regulator, frequently mutated in UC, could affect metformin response;
7. Phosphatase and tensin homolog (PTEN) staining

   Cell cycle regulator, frequently inactivated in invasive UC, affects metformin response;
8. p53 staining

Tertiary Endpoints The following parameters will be investigated through the analysis of any differences in either their values between the time of enrollment and the day of surgery or differences in the frequency between the treatment and control groups.

Between time of enrollment and date of surgery;

1. Serum Insulin
2. Fasting glucose levels
3. Body mass index
4. Changes in serum prostate specific antigen (PSA)

   Clinical Marker of efficacy, has been shown to affect prognosis:
5. Pathologic T0 rate at cystectomy vs. historical rates

   Potential Novel Biomarkers:
6. Number of circulating tumor cells or tumor microparticles before and after treatment with metformin

   The following additional stratification analyses of the data will be performed in order to assess our results in light of prior research findings:

   Stratification of Pathologic Markers;
7. Stratification of pAKT and Survivin expression levels by the presence or absence of PTEN expression
8. Stratification of TUNEL and Ki67 by the status of p53 staining
9. Stratification of pathologic markers by the use or absence of administration of neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years and 85≤.
2. Patients must have biopsy proven invasive bladder cancer by TURBT, previously untreated prior to TURBT by systemic chemotherapy.
3. Patients must be able to swallow and tolerate oral medication
4. Hemoglobin A1c ≤ 6.5%.
5. Able to comprehend written and verbal study instructions related to study protocol and provide informed consent.
6. Any women with childbearing potential must use a highly effective contraception method, of which include: hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation.

Exclusion Criteria

1. Patient has been treated for a prior cancer diagnosis with cisplatin-derived chemotherapy regimens or has had pelvic radiation therapy.
2. Previous or current diagnosis of type 1 or 2 diabetes mellitus.
3. Metformin exposure within the previous 12 months.
4. Expected or simultaneous use of sulfonylureas, thiazolidinediones, or insulin.
5. Known metformin allergy or intolerance.
6. Participation in another drug trial either within 30 days prior to study enrollment or during the time when they are on study protocol.
7. Serious cardiovascular disease including myocardial infarction within 6 months, unstable angina, serious cardiac arrythmias excluding atrial fribrillation, or cerebrovascular accident within 6 months prior to screening visit.
8. Abnormal liver function tests: Total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) > 1.8 X upper limit of normal
9. Estimated glomerular filtration rate (eGFR) of ≤40 mL/min.
10. History of other malignancy, except non-muscle invasive bladder cancer, treated non-melanoma skin cancer, stage I melanoma and solid tumors adequately treated, with no persistent evidence of disease for 5 years.
11. Concomitant medical condition predisposing to metformin hydrochloride-associated lactic acidosis; examples include NYHA class III or IV congestive heart failure, history of acidosis and chronic alcohol intake averaging ≥ 4 beverages per day.
12. A history of rhabdomyolysis.
13. The use of medications including niacin and colchicine, as well as strong inhibitors of cytochrome p-450 3A4 (see list in section 4.2).
14. Untreated hypothyroidism.
15. Pregnancy.
16. Breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Bladder tumor proliferation rate | The participant will be followed for the duration of the pre-surgical preparation period. This is expected to be fewer than 12 weeks
  The primary endpoint of this trial will be the assessment of the tumor proliferation rate. This will be investigated through the analysis of the change in Ki67 (cellular marker of cell proliferation) tissue staining between the TURBT tissue samples and the cystectomy tissue.
Feasibility of performing neoadjuvant window of opportunity trials using drugs with potential bioactivity against invasive bladder cancer | The participant will be followed for the duration of the pre-surgical preparation period. This is expected to be fewer than 12 weeks
  This trial is also designed to establish the framework and evaluate the feasibility of performing neoadjuvant window of opportunity trials using drugs with potential bioactivity against invasive bladder cancer at the London Health Sciences Center. The goal is to accrue 44 patients within 18 months to the trial, and the study will be prematurely closed if fewer than 10 patients are recruited within 12 months.

SECONDARY OUTCOMES:
Toxicity in patients who participate in the treatment regimen of Metformin and Simvastatin therapy | The participant will be followed for the duration of the pre-surgical preparation period. This is expected to be fewer than 12 weeks
  This study will assess the rate of grade 3 or higher toxicity caused by the study drug combination as defined by the CTCAE 4.03.
Level of apoptosis observed in tumor cells of patients who undergo Metformin and Simvastatin therapy before cystectomy. | The participant will be followed for the duration of the pre-surgical preparation period. This is expected to be fewer than 12 weeks
  Tissue will be analyzed for the change in the marker of apoptosis Terminal deoxynucleotidyl Transferase-mediated dUTP nick end labeling (TUNEL) staining between TURBT and cystectomy tissue samples.
Impact of Metformin and Simvastatin therapy on the signalling pathways involved in invasive urothelial carcinoma. | The participant will be followed for the duration of the pre-surgical preparation period. This is expected to be fewer than 12 weeks
  Various signalling pathways involved in cell proliferation and metformin response that may be affected by the combination of study drugs will be evaluated by analyzing tissue samples obtained from the patient during TURBT and then cystectomy. These experiments will be done to assess whether the combination of study drugs are able to inhibit the cellular signalling pathways that contribute to cancer cell growth by comparing the signaling levels between pre and post treatment samples. These pathways include PI3K/Akt/mTOR and AMPK. We will also evaluate the effect of the levels of PTEN and p53 on the cell response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Izawa, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Center; Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No